CLINICAL TRIAL: NCT03265210
Title: "Relief": A Behavioral Intervention for Depression and Chronic Pain in Primary Care
Brief Title: A Behavioral Intervention for Depression and Chronic Pain in Primary Care
Acronym: Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1704018104; 5P50MH113838 (NIH)
Record Dates: First submitted 2017-08-10; First posted 2017-08-29 (Actual); Results first posted 2023-02-24 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Chronic Pain; Depression
Keywords: Middle-aged and Older Adults; Primary Care
MeSH Terms: conditions — Chronic Pain; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research assistants will be blind to who is receiving Relief and who is not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relief (Experimental): Relief relies on a neurobiological model to simplify its behavioral targets and uses mobile technology to augment its interventions. Relief was co-developed with our primary care partners with the goal to be usable by non-physician clinicians of primary care offices eligible to provide billable services.
  Interventions: Behavioral: RELIEF
- Referral (No Intervention): Referral for mental health based on clinical indication.

INTERVENTIONS:
Behavioral: RELIEF — A 9-week behavioral intervention for primary care designed to reduce depression and pain-related disability.
  Arms: Relief

SUMMARY:
Chronic pain and depression frequently co-exist in late and mid-life and contribute to increased disability, high health care costs, psychiatric comorbidity, and suicide. The investigators will recruit 60 adults from Weill Cornell Medical Associates primary care practices; participants will be randomized to either Relief (a 9 session behavioral intervention) or usual care/referral for mental health care. Research assessments are conducted with both groups at study entry (Baseline), 6, 9, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years
* PHQ-9 greater than or equal to 10
* Non-cancer related chronic pain, defined as pain during most days over the past 3 months by patient report
* Capacity to consent

Exclusion Criteria:

* DSM-5 Axis 1 other than depression and anxiety disorders
* Montreal Cognitive Assessment (MoCA) < 24
* Active suicidal ideation, i.e. MADRS Suicide Item greater than or equal to 4
* Severe or life-threatening medical illness.
* Patients on psychotropics, opioids or benzodiazepines will be included if they do not meet DSM-5 criteria for opioid, anxiolytics or other substance abuse disorders

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Kiosses, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - Weill Cornell Internal Medicine Associates (WCIMA), New York, New York
  - Iris Cantor Men's & Women's Health Centers, New York, New York
  - Irving Sherwood Wright Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this study is submitted to the National Database for Clinical Trials related to Mental Illness (NDCT). The NDCT is run by NIH and allows researchers studying mental health to collect and share information with each other. Researchers must apply to NIH in order to be allowed access to the data for 1 year's time; after which they must re-apply.
Time Frame: Data will be available as per NIH's data sharing policy.
Access Criteria: Access criteria is determined by NIH and can be requested by applying online.
URL: https://nda.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Relief | Referral
Started | 50 | 23
Completed | 38 | 14
Not Completed | 12 | 9
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Relief | Referral | Total
Number analyzed (Participants) | 50 | 23 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.28 (10.09) | 68.65 (10.72) | 67.71 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 17 | 56
  Male | 11 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 44 | 19 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 5 | 21
  White | 32 | 14 | 46
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 50 | 23 | 73

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinically Significant Depressive Symptoms, as Measured by the Montgomery Asberg Depression Rating Scale (MADRS)
Description: The MADRS is a 10 item questionnaire assessing severity of depression by scoring participants on mood, anxiety, sleep, concentration, appetite, and suicidal thoughts. The lowest score is 0, no depression symptoms, and the highest possible score is 60, severe depression symptoms.
Time Frame: Baseline, 6, 9, and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relief | Referral
Number analyzed (Participants) | 50 | 23
score on a scale
  Baseline Totals | 19.37 (7.27) | 20.87 (5.85)
  Week 6 Totals | 14.88 (6.73) | 18.67 (6.88)
  Week 9 Totals | 16.44 (7.66) | 18.00 (7.51)
  Week 12 Totals | 13.30 (7.39) | 16.67 (6.97)
Statistical Analysis 1: Comparison: Relief vs Referral; Baseline; Test type: Superiority; p = 0.39, t-test, 2 sided; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-4.95 to 1.95] — Mean value in Relief Arm minus Mean value in Referral Arm
Statistical Analysis 2: Comparison: Relief vs Referral; 6 weeks; Test type: Superiority; p = 0.03, t-test, 2 sided; Mean Difference (Final Values) = -3.79, 95% CI 2-sided [-7.19 to -0.39] — Mean value in Relief Arm minus Mean value in Referral Arm
Statistical Analysis 3: Comparison: Relief vs Referral; 9 weeks; Test type: Superiority; p = 0.42, t-test, 2 sided; Mean Difference (Final Values) = -1.56, 95% CI 2-sided [-5.38 to 2.26] — Mean value in Relief Arm minus Mean value in Referral Arm
Statistical Analysis 4: Comparison: Relief vs Referral; 12 weeks; Test type: Superiority; p = 0.07, t-test, 2 sided; Mean Difference (Final Values) = -3.37, 95% CI 2-sided [-7.02 to 0.28] — Mean value in Relief Arm minus Mean value in Referral Arm

2. Primary Outcome: Change in Pain-related Disability, as Measured by the Roland-Morris Disability Questionnaire (RMDQ)
Description: The RMDQ includes a scale assessing how much pain the participant has experienced in the past week, with 0 indicating no pain and 10 indicating pain as bad as he/she can imagine; scores will be listed under domain 1. In addition, the RMDQ also includes a series of questions related to pain disability, with 0 indicating no pain-related disability, and 24 indicating severe pain-related disability; scores will be listed under domain 2.
Time Frame: Baseline, 6, 9, and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relief | Referral
Number analyzed (Participants) | 50 | 23
score on a scale
  Domain 1: Baseline | 5.83 (2.09) | 6.57 (2.21)
  Domain 1: Week 6 | 5.85 (2.23) | 6.47 (1.81)
  Domain 1: Week 9 | 5.54 (2.75) | 6.60 (1.59)
  Domain 1: Week 12 | 5.58 (2.38) | 6.67 (1.72)
  Domain 2: Baseline | 13.17 (5.25) | 16.36 (5.72)
  Domain 2: Week 6 | 11.70 (5.24) | 16.00 (6.02)
  Domain 2: Week 9 | 10.26 (5.59) | 16.21 (6.15)
  Domain 2: Week 12 | 11.05 (6.20) | 15.40 (6.20)
Statistical Analysis 1: Comparison: Relief vs Referral; Domain 1, Baseline; Test type: Superiority; p = 0.17, t-test, 2 sided; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-1.81 to 0.33] — Mean value in Relief Arm minus Mean value in Referral Arm
Statistical Analysis 2: Comparison: Relief vs Referral; Domain 1, 6 weeks; Test type: Superiority; p = 0.25, t-test, 2 sided; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-1.68 to 0.44] — Mean value in Relief Arm minus Mean value in Referral Arm
Statistical Analysis 3: Comparison: Relief vs Referral; Domain 1, 9 weeks; Test type: Superiority; p = 0.09, t-test, 2 sided; Mean Difference (Final Values) = -1.06, 95% CI 2-sided [-2.29 to 0.17] — Mean value in Relief Arm minus Mean value in Referral Arm
Statistical Analysis 4: Comparison: Relief vs Referral; Domain 1, 12 weeks; Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = -1.09, 95% CI 2-sided [-2.19 to 0.01] — Mean value in Relief Arm minus Mean value in Referral Arm
Statistical Analysis 5: Comparison: Relief vs Referral; Domain 2, Baseline; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Final Values) = -3.19, 95% CI 2-sided [-5.90 to -0.48] — Mean value in Relief Arm minus Mean value in Referral Arm
Statistical Analysis 6: Comparison: Relief vs Referral; Domain 2, 6 weeks; Test type: Superiority; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-7.06 to -1.54] — Mean value in Relief Arm minus Mean value in Referral Arm
Statistical Analysis 7: Comparison: Relief vs Referral; Domain 2, 9 weeks; Test type: Superiority; p = 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -5.95, 95% CI 2-sided [-8.85 to -3.05] — Mean value in Relief Arm minus Mean value in Referral Arm
Statistical Analysis 8: Comparison: Relief vs Referral; Domain 2, 12 weeks; Test type: Superiority; p = 0.007, t-test, 2 sided; Mean Difference (Final Values) = -4.35, 95% CI 2-sided [-7.46 to -1.24] — Mean value in Relief Arm minus Mean value in Referral Arm

3. Primary Outcome: Client Satisfaction Questionnaire (CSQ)
Description: A questionnaire that evaluates participants' satisfaction with treatment; ranging from 1 (needs have not been met/dissatisfied) to 4 (almost all needs have been met/very satisfied).
  Domain 1 measures met needs. Scores range from 0-4 and higher scores indicate more needs met. Domain 2 measures satisfaction with services. Scores range from 0-4 and higher scores indicate more satisfaction with services. Domain 3 measures willingness to return. Scores range from 0-4 and higher scores indicate greater willingness to return.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relief | Referral
Number analyzed (Participants) | 50 | 23
score on a scale
  Domain 1 | 3.40 (0.81) | 2.29 (1.70)
  Domain 2 | 3.72 (0.51) | 3.20 (0.79)
  Domain 3 | 3.67 (0.68) | 2.71 (1.89)
Statistical Analysis 1: Comparison: Relief vs Referral; Domain 1; Test type: Superiority; p = 0.0003, t-test, 2 sided; Mean Difference (Final Values) = 1.11, 95% CI 2-sided [0.53 to 1.69] — Mean value in Relief Arm minus Mean value in Referral Arm
Statistical Analysis 2: Comparison: Relief vs Referral; Domain 2; Test type: Superiority; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [0.21 to 0.83] — Mean value in Relief Arm minus Mean value in Referral Arm
Statistical Analysis 3: Comparison: Relief vs Referral; Domain 3; Test type: Superiority; p = 0.002, t-test, 2 sided; Mean Difference (Final Values) = 0.96, 95% CI 2-sided [0.36 to 1.56] — Mean value in Relief Arm minus Mean value in Referral Arm

4. Secondary Outcome: Change in Mood, as Measured by the Daily Photographic Affect Meter (PAM)
Description: The PAM is used for assessing mood and emotional state. Participants can either score a "positive" or "negative" affect value. PAM uses photos that user selects and map it to arousal (y-axis) and valence(x-axis). Domain 1 is derived from PAM using y-axis (column score): (low activation to high activation): takes on discrete values ranging from 1 - 5. Domain 2 is derived from PAM using x-axis (row score): (unpleasurable to pleasurable or negative to positive): takes on discrete values ranging from 1 - 4.
Time Frame: Daily for 12 weeks
Population: Data was extracted from wearable devices worn by study participants. Once data was retrieved, some passively collected data was filtered and patients with invalid data points were removed as per study biostatistician.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relief | Referral
Number analyzed (Participants) | 18 | 2
score on a scale
  Domain 1 | 2.83 (1.02) | 2.48 (1.01)
  Domain 2 | 2.58 (0.96) | 2.94 (0.84)

5. Secondary Outcome: Activities Monitoring
Description: Activities monitoring through a phone application; measuring distance in meters covered daily by the participant during the week.
Time Frame: Daily for 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Relief | Referral
Number analyzed (Participants) | 18 | 2
meters | 20085.61 (174446.40) | 1654.16 (4581.61)

6. Secondary Outcome: Activities Monitoring
Description: Activities monitoring through a phone application; measuring number of places visited daily during the week. Data is based on the total uptime of the location stream (unit is continuous seconds).
Time Frame: Daily for 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Relief | Referral
Number analyzed (Participants) | 18 | 2
seconds | 75947.60 (23672.34) | 69557.39 (29401.19)

ADVERSE EVENTS:
Time Frame: 12 weeks (total duration of study)
Arm/Group | Relief | Referral
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/23
Serious Adverse Events (participants affected / at risk) | 4/50 | 0/23
Other Adverse Events (participants affected / at risk) | 3/50 | 1/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relief (N=50) | Referral (N=23)
Hospitalization (Cardiac disorders) | 2 (2) | 0 (0) — Participant admitted to hospital for atrial fibrillation. Participant admitted to hospital for tachycardia following radiation treatment.
Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) — Participant psychiatrically hospitalized.
Surgery (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Participant had scheduled surgery to remove tumor on lung.
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Participant hospitalized for numbness and dysphagia following treatment for esophageal cancer.
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relief (N=50) | Referral (N=23)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) — Participants experienced rash on wrist underneath study smart watch. No medical attention necessary; went away on its own.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT03265210/Prot_002.pdf
  • Statistical Analysis Plan (2016-10-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT03265210/SAP_003.pdf